CLINICAL TRIAL: NCT03562130
Title: A Monocentric Single-arm Study to Characterize the Long-term Safety, Efficacy, and Pharmacodynamic of GLP-2 Analog (Revestive®) in the Management of Short Bowel Syndrome Pediatric Patients on Home-parenteral Nutrition (HPN)
Brief Title: Characterization of the Long-term Safety, Efficacy, and Pharmacodynamics Revestive® in the Management of Short Bowel Syndrome Pediatric Patients
Acronym: REVE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Imagine Institute (Other); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P171002J; 2017-001405-32 (EudraCT Number)
Record Dates: First submitted 2018-05-18; First posted 2018-06-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Short Bowel Syndrome
Keywords: Teduglutide; Short Bowel Syndrome; Parenteral nutrition; Intestinal failure
MeSH Terms: conditions — Short Bowel Syndrome; Hyperphagia; Intestinal Failure | interventions — teduglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Revestive (Experimental): Revestive® (teduglutide)is administered in children sub cutaneous injection at 0.05 mg/kg body weight once daily
  Interventions: Drug: Teduglutide

INTERVENTIONS:
Drug: Teduglutide — Daily sub cutaneous injection 0,05 mg/kg/day

SUMMARY:
The purpose of this study is to evaluate if the treatment could maximize intestinal absorption, minimize the inconvenience of diarrhea, and avoid, reduce or eliminate the need for parenteral support (PS) to achieve normal growth, to avoid parenteral nutrition complications and to achieve the best possible quality of life for the patient

DETAILED DESCRIPTION:
The short bowel syndrome (SBS) may be defined as a severe malabsorption caused by reduction of intestinal absorptive surface following massive resection of the small intestine. Teduglutide (Revestive®) is an analog of glucagon-like peptide 2 (GLP-2), a naturally occurring hormone that regulates the functional and structural integrity of the cells lining the gastrointestinal tract. The aim of the treatment is to maximize intestinal absorption, minimize the inconvenience of diarrhea, and avoid, reduce or eliminate the need for parenteral support (PS) to achieve the best possible quality of life for the patient. The rationale for the use of Revestive® is based on data obtained, especially in the trial in SBS patients.

Treatment with 0.05 mg/kg/day was safe and well tolerated (no recorded side effects).

Patients remained stable despite substantial reduction in parenteral nutrition (PN) supply as evidenced by stable body weight and height, serum electrolytes, pancreatic enzymes and renal function tests.

Treatment was associated with:

* Reduced PN volume and calories delivered by 25 and 45% respectively with 20% of patients weaned off PN during the study period
* Increased Enteral Nutrition (EN) supply in volume and calories by 40 and 62% respectively
* Increased in plasma citrulline during the treatment period, but decreased after Teduglutide discontinuation The recommended dose of Revestive® in children and adolescents (aged 1 to 17 years) is the same as for adults (0.05 mg/kg body weight once daily).

ELIGIBILITY:
Inclusion Criteria:

* Being aged from 2 to 18 years old included ;
* Presenting less than 80 cm of residual small intestine with or without the terminal ileum, ileocecal valve and right colon or having less than 120 cm in case of Short Bowel Syndrome (SBS) caused by Hirschsprung disease;
* Being stable on PN support (inability to significantly reduce PN intake for the last six months before inclusion) ;
* Being dependent on PN for at least 2 years and enterally fed (oral or tube feeding) ;
* Having a normal colonoscopy in the 12 months before screening for children with maintained colon (=SBS type 2 or 3) older than 12 years ;
* Having signed the Informed consent form (or parents or legal representative for minor patients).

Exclusion Criteria:

* Having a major gastrointestinal surgical intervention like serial transverse enteroplasty or any other bowel lengthening procedure performed within 6 months of screening ;
* Having a clinically significant untreated intestinal obstruction or active stenosis ;
* Having an unstable absorption due to cystic fibrosis or known DNA abnormalities ;
* Presenting a radiographic or manometric evidence of pseudo-obstruction or severe known dysmotility syndrome, including persistent, severe gastroschisis-related motility disorders ;
* Having an unstable cardiac disease, congenital heart disease or cyanotic disease, with the exception of patients who had undergone ventricular or atrial septal defect repair ;
* Having a history of cancer or clinically significant lymphoproliferative disease; excepted resected cutaneous basal or squamous cell carcinoma, or in situ non-aggressive and surgically resected cancer ;
* Having participated in a clinical study using an experimental drug within 1 month or an experimental antibody treatment within 3 months prior to screening, or concurrent participation in any clinical study using an experimental drug that would affect the safety of teduglutide ;
* Having already used native GLP-2 and glucagon-like peptide-1 analog or human growth hormone within 3 months prior to screening ;
* Having already used oral or IV glutamine, octreotide, or dipeptidyl peptidase IV (DPP-IV) inhibitors within 3 months prior to screening ;
* Having an active Crohn's disease which has been treated with biological therapy within the 6 months prior to screening ;
* Having an intestinal polyposis;
* Being, for female patient, both lactating and breast-feeding or having a positive pregnancy test during the screening period;
* Refusing the follow the protocol requirements in terms of birth control ;
* Being unable to follow the study procedures for any reason: psychological, geographical…
* Hypersensitivity to the active substance or to any of the excipients listed in section 6.1 of Summary of Product Characteristics (SPC), or trace residues of tetracycline.
* Active or suspected malignancy.
* Patients with a history of malignancies in the gastrointestinal tract including the hepatobiliary system within the last five years.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Decrease in parenteral nutrition: Parenteral Nutrition/Resting Energy Expenditure (PN/REE) | At week 24
  Evaluate the efficacy of Revestive® treatment

SECONDARY OUTCOMES:
Ostomy output defined as stool balance testing, urine output and plasma citrulline | up to week 48
  Evaluate the impact of Revestive on ostomy flow
Change in days per week of Parenteral Nutrition (PN) | up to week 48
  Quantify the impact of Revestive on the number of perfusion in a week
Change in number of stool per day | up to week 48
  to evaluate the impact of Revestive on diarrhea
Change in stools consistency (Bristol stool chart) | up to week 48
  to evaluate the impact of Revestive on diarrhea
Ingesta (calorimetric measure) | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Stool weight/24h | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Percentage of lipid in stool | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Percentage of nitrogen in stool | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Percentage of carbohydrate in stool | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Percentage of sodium in stool | Every 4 weeks up to week 48
  to evaluate the impact of Revestive on Intestinal absorption
Number of adverse events | At week 48
  to evaluate the long term safety of Revestive
Change in body weight | At baseline, then at 6 and 12 months
Change in heart rate | At baseline, then at 6 and 12 months
Change in blood pressure | At baseline, then at 6 and 12 months
Endogenous GLP-2 rates (antibody ELISA) | up to week 48
  to evaluate the response rate of Revestive

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GOULET, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker - Enfants malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lambe C, Talbotec C, Kapel N, Barbot-Trystram L, Brabant S, Nader EA, Pigneur B, Payen E, Goulet O. Long-term treatment with teduglutide: a 48-week open-label single-center clinical trial in children with short bowel syndrome. Am J Clin Nutr. 2023 Jun;117(6):1152-1163. doi: 10.1016/j.ajcnut.2023.02.019. Epub 2023 May 3. PMID 37270289